CLINICAL TRIAL: NCT01637116
Title: Profiling Urticaria for the Identification of Subtypes
Acronym: PURIST
Status: Completed | Type: Observational
Sponsor: Marcus Maurer (Other)
Responsible Party: Sponsor-Investigator, Marcus Maurer, Professor, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: PURIST
Record Dates: First submitted 2011-08-15; First posted 2012-07-10 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Non-autoreactive Chronic Spontaneous Urticaria; Autoimmune Chronic Spontaneous Urticaria; Autoreactive, Non-autoimmune Chronic Spontaneous Urticaria

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- autoimmune chronic spontaneous urticaria: Patients with chronic spontaneous urticaria with a positive ASST, who also test positive in a cell activating assay (BHRA OR CD 63 activation of healthy donor basophils) and who exhibit anti-FcεRI and/or anti-IgE autoantibodies (=autoimmune chronic spontaneous urticaria).
- autoreactive, non-autoimmune chronic spontaneous urticaria: Patients with chronic spontaneous urticaria with a positive ASST, who test negative in cell activation assay or who do not exhibit anti-FcεRI or anti-IgE autoantibodies (=autoreactive, non-autoimmune chronic spontaneous urticaria)
- non-autoreactive chronic spontaneous urticaria: Patients with chronic spontaneous urticaria and a negative ASST (= non-autoreactive chronic spontaneous urticaria)

SUMMARY:
The primary purpose of this study is to identify and characterize novel diagnostic markers for autoimmune urticaria, a subset of chronic spontaneous urticaria.

Additional aims: include the comparison of the clinical profiles of autoreactive, autoimmune and non autoreactive / autoimmune urticaria and the quality of life impairment in these subsets of chronic spontaneous urticaria.

ELIGIBILITY:
Inclusion Criteria:

* chronic spontaneous urticaria
* disease duration > 6 weeks
* signed and dated informed consent
* age 18 years or older
* Non sedating antihistamines may be used on an "on demand" basis throughout the study, in case of high urticaria activity [>50 wheals, and intense pruritus: urticaria activity score (UAS) of 6] or in case of an emergency. Patients may take either cetirizine 10 mg up to a maximum of 4 tablets per 24 hours or fexofenadine 180 mg up to a maximum of 4 tablets per 24 hours. The use of antihistamines and the reason has to be documented by the patient in the patient diary. Patients should avoid the use of antihistamines during the study and especially during the three days prior to skin testing
* for female with childbearing potential: female will have to use a safe method of contraception to prevent pregnancy and will have to agree to continue this method of contraception during the whole study.

Exclusion Criteria:

* intake of immunosuppressives 3 month before Screening Visit and during the course of the study. Immunosuppressives including ciclosporin, methotrexate, mycophenolate, azathioprine and cyclophosphamide need to be stopped at least 3 month before Screening Visit
* intake of corticosteroids (e.g. oral, injection) 1 month before Screening Visit and during the course of the study. Corticosteroids need to be stopped at least 1 month before the Screening Visit.
* Previous or present treatment with anti-IgE-antibodies including omalizumab (Xolair)
* age below 18 years
* use of tricyclic antidepressants (e.g. amitriptyline), doxepin, leukotriene antagonists (e.g. montelukast, trade name: singulair), H2 antihistamines (e.g. cimetidine, famotidine, ranitidine), sulphasalazine, dapsone, tranexamic acid, warfarin, heparin during the last 4 weeks before the Screening Visit and during the course of the study.
* pregnancy, lactation or planned pregnancy during the study
* mentally incapacitated subjects
* patients protected by the law (adults under guardianship, or hospitalized in a public or private institution for a reason other than the study, or incarcerated)
* patients suffering from urticaria vasculitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with chronic spontaneous urticaria and a negative ASST (= non-autoreactive chronic spontaneous urticaria)
  2. Patients with chronic spontaneous urticaria with a positive ASST, who also test positive in a cell activating assay (BHRA OR CD 63 activation of healthy donor basophils) and who exhibit anti-FcεRI and/or anti-IgE autoantibodies (=autoimmune chronic spontaneous urticaria).
  3. Patients with chronic spontaneous urticaria with a positive ASST, who test negative in cell activation assay or who do not exhibit anti-FcεRI or anti-IgE autoantibodies (=autoreactive, non-autoimmune chronic spontaneous urticaria)
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2011-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Results of the ASST | 21 days per patient
  to identify and characterize novel diagnostic markers for autoimmune urticaria, a subset of chronic spontaneous urticaria
Results of a cell activating assay (BHRA) | 21 days per patient
  to identify and characterize novel diagnostic markers for autoimmune urticaria, a subset of chronic spontaneous urticaria
Results of autoantibody-test (anti-IgE and anti-FcRI) | 21 days per patient
  to identify and characterize novel diagnostic markers for autoimmune urticaria, a subset of chronic spontaneous urticaria

SECONDARY OUTCOMES:
Results of Urticaria activity score (UAS7) | 21 days per patient
  comparison of the clinical profiles of autoreactive, autoimmune and non autoreactive / autoimmune urticaria and the quality of life impairment in these subsets of chronic spontaneous urticaria
Results of HRQoL scores (CU-Q2oL, DLQI) | 21 days per patient
  comparison of the clinical profiles of autoreactive, autoimmune and non autoreactive / autoimmune urticaria and the quality of life impairment in these subsets of chronic spontaneous urticaria
Results of laboratory tests (Thyroid antibodies (anti-TPO +/- anti-thyreoglobulin); ANA; Rheumatoid factor; CRP; ESR; total IgE; T3,T4, TSH, diff BB, Helicobacter pylori stool antigen test or breath test; D-Dimer) | 21 days per patient
  comparison of the clinical profiles of autoreactive, autoimmune and non autoreactive / autoimmune urticaria and the quality of life impairment in these subsets of chronic spontaneous urticaria

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Maurer, Prof. Dr. med., Principal Investigator — Charite-Universitätsmedizin Berlin
Locations (1):
- University of Berlin Charité, Berlin, State of Berlin, Germany